CLINICAL TRIAL: NCT04676984
Title: Medication Use and Quality of Life Among Older People (Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Carina Lundby, Postdoctoral Researcher, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ODIN-1 Pilot
Record Dates: First submitted 2020-12-01; First posted 2020-12-21 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Reduction, Harm
Keywords: Deprescribing; Polypharmacy; Guideline
MeSH Terms: conditions — Harm Reduction | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consultations (Other): The intervention will comprise a series of consultations between the patient and general practitioner (at least three), where the patient and general practitioner will continuously adjust the patient's medication according to the patient's goals, needs, and preferences.
  Interventions: Other: Consultations

INTERVENTIONS:
Other: Consultations — The intervention will comprise a series of consultations between the patient and general practitioner (at least three), where the patient and general practitioner will continuously adjust the patient's medication according to the patient's goals, needs, and preferences.

SUMMARY:
This project will provide new evidence on how to optimize medication use among older people with limited life expectancy. This will be done by testing whether a patient-centered deprescribing intervention, focused on aligning medical treatment with patients' preferences, can improve quality of life among older people with limited life expectancy. This registration concerns the initial pilot study.

DETAILED DESCRIPTION:
In a pragmatic randomized controlled trial, this project will test whether a comprehensive and patient-centered deprescribing intervention can improve quality of life among older people with limited life expectancy. This registration concerns the initial pilot study. All patients included in the pilot study will receive the intervention (that is, the pilot study will not include randomization).

The intervention will comprise a series of consultations between the patient and general practitioner (GP) (at least three) to continuously adjust the patient's medication according to the patient's goals, needs, and preferences, thereby ensuring alignment with the patient's priorities. Thus, the purpose of this intervention is to initiate and facilitate a continued deprescribing process. The process can be summarized in seven steps: During an initial consultation (1: Consultation 0), the GP assesses patient eligibility. If the patient would like to participate, a project nurse subsequently visits the patient at home (2: Home visit) for retrieval of informed consent as well as baseline measurements. During the next consultation (3: Consultation 1), the patient and GP discuss how the patient feels about his/her medical treatment, and the GP provides the patient with written material for the patient to prepare prior to the next consultation. The patients prepares (4: Preparation) by considering and verbalizing his/her goals of care and treatment preferences. Simultaneously, a clinical pharmacist examines the patient's medication list and provides suggestions to the GP on which drugs can be continued and deprescribed, respectively. During the next consultation (5: Consultation 2), the patient and GP discuss the patient's preferences and initiate deprescribing initiatives aligned with the patient's priorities. During a new consultation (6: Consultation 3), the patient and GP follow up on the changes initiated and initiate new deprescribing initiatives if such can be identified. If needed, subsequent consultations (7: Consultation X) are planned until the patient and GP consider the patient's medical treatment optimal.

ELIGIBILITY:
Inclusion criteria:

* Aged ≥80 years
* Take ≥8 different medications
* Have a life expectancy of <2 years, estimated via the Surprise Question ("Would you be surprised if this patient died within 1-2 years?") by the general practitioner
* Have a Mini-Mental State Exam (MMSE) score of ≥15
* Are able to provide informed consent

Exclusion Criteria:

* Not able to communicate
* Does not speak and understand Danish

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
HEALTH-RELATED QUALITY OF LIFE | Baseline
  Health-related quality of life will be measured using the Danish version of the SF-12v2 Health Survey.
CHANGE FROM BASELINE HEALTH-RELATED QUALITY OF LIFE AT 3 MONTHS | 3 months
  Health-related quality of life will be measured using the Danish version of the SF-12v2 Health Survey.
CHANGE FROM BASELINE HEALTH-RELATED QUALITY OF LIFE AT 6 MONTHS | 6 months
  Health-related quality of life will be measured using the Danish version of the SF-12v2 Health Survey.
HEALTH-RELATED QUALITY OF LIFE (DEPRESSION) | Baseline
  Health-related quality of life will be measured using the Danish version of the Depression List.
CHANGE FROM BASELINE HEALTH-RELATED QUALITY OF LIFE (DEPRESSION) AT 3 MONTHS | 3 months
  Health-related quality of life will be measured using the Danish version of the Depression List.
CHANGE FROM BASELINE HEALTH-RELATED QUALITY OF LIFE (DEPRESSION) AT 6 MONTHS | 6 months
  Health-related quality of life will be measured using the Danish version of the Depression List.
MORTALITY | 3 months
  Mortality will be assessed through the nationwide Danish Central Person Registry.
MORTALITY | 6 months
  Mortality will be assessed through the nationwide Danish Central Person Registry.
MORTALITY | 12 months
  Mortality will be assessed through the nationwide Danish Central Person Registry.

SECONDARY OUTCOMES:
COGNITIVE FUNCTION | Baseline, 3 months and 6 months
  Cognitive function will be measured using the Danish version of the Mini-Mental State Examination-2 (MMSE-2) Standard Form.
FUNCTIONAL LEVEL | Baseline, 3 months and 6 months
  Functional level will be measured using the Danish version of the Vulnerable Elders Survey 13 (VES-13).
HAND-GRIP STRENGTH | Baseline, 3 months and 6 months
  Hand-grip strength will be measured using a hand-grip dynamometer.
ABILITY TO SIT AND STAND | Baseline, 3 months and 6 months
  Ability to sit and stand will be measured via the 30-second stand-sit-test.
NUMBER OF MEDICATIONS DISCONTINUED | 3 months, 6 months and 12 months
  Number of medications dicontinued will be assessed through the medication lists.
NUMBER OF MEDICATION CHANGES | 3 months, 6 months and 12 months
  Number of medication changes will be assessed through the medication lists.
HOSPITAL ADMISSIONS | 3 months, 6 months and 12 months
  Admissions will be assessed through the nationwide Danish National Patient Register.
HEALTH CARE COSTS | 3 months, 6 months and 12 months
  Health care costs.
SUCCESS RATE OF THE INTERVENTION | 3 months, 6 months and 12 months
  Succes rate of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Pottegård, Prof, Principal Investigator — apottegaard@health.sdu.dk
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No